CLINICAL TRIAL: NCT05674552
Title: Efficacy of Exogenous Ketone Esters for Children With Refractory Convulsive Status Epileptics
Brief Title: Exogenous Ketone Esters for Refractory Status Epileptics
Acronym: EKERSE
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Elsayed Abdelkreem, Lecturer of Pediatrics, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-22-12-46
Record Dates: First submitted 2022-12-18; First posted 2023-01-06 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Status Epilepticus
Keywords: Status epilepticus; Refractory status epilepticus; Generalized convulsive status epilepticus; Exogenous ketone esters; Children; Seizures
MeSH Terms: conditions — Status Epilepticus; Seizures

STUDY DESIGN:
Intervention Model Description: Eligible children will be randomized into two equal-sized groups. Study group: will receive exogenous ketone esters plus standard of care. Control group: will receive only standard of care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Children receiving exogenous ketone esters + standard of care
  Interventions: Drug: Exogenous ketone ester
- Control group (No Intervention): Children receiving only standard of care

INTERVENTIONS:
Drug: Exogenous ketone ester — 500 mg/kg over 5 min administered by nasogastric tube, followed after 1 hr by repeated hourly doses of 125 mg/kg for 8 hrs.
  Arms: Study group

SUMMARY:
This study aims to investigate the efficacy of add-on exogenous ketone esters for the treatment of children with refractory generalized convulsive status epilepticus

DETAILED DESCRIPTION:
Generalized convulsive status epilepticus (GCSE) is a common neurological emergency in children with significant morbidity and mortality. Benzodiazepines (Bzs) are the initial anti-seizure medications (ASMs) for children with GCSE, but nearly a third of cases are not controlled by (Bzs). Moreover, about 40% of cases not responding to BZs are not controlled by second-line ASMs.

Ketogenic diet (KD) has been classically used for treating children with drug resistant epilepsy. Recently, KD has been used for refractory and super refractory status epilepticus. However, KD takes time to achieve ketosis and may be practically challenging in emergency situations and critically ill patients. Exogenous ketone esters (EKE) could be a more convenient and rapid way to achieve ketosis in acute settings.

ELIGIBILITY:
Inclusion Criteria:

* Refractory Generalized convulsive status epilepticus.

Exclusion Criteria:

* Failure to obtain informed consent.
* Recent intake of exogenous ketones, ketogenic diet, or any dietary restrictions/modifications.
* Hemodynamic or cardio-respiratory instability.
* Traumatic brain injury.
* Hypo-/hyperglycemia.
* Metabolic acidosis.
* Ketosis (βHB > 2 mmol/L).
* Associated severe disease condition, including hepatic, renal, respiratory, cardiac, gastrointestinal, endocrinal, and immune systems.
* Malnutrition/obesity.
* Limitations to nasogastric tube feeding.
* Inborn errors of metabolism.
* Allergies or any other contraindication to exogenous ketone esters.
* Current or recent (within the last 24 hours) propofol therapy.
* Intake of carbonic-anhydrase inhibitors.

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving electroclinical cessation of seizures | 60 minutes
  Proportions of patients who achieve cessation of BOTH clinical seizures (as observed clinically) AND electrical seizures (evaluated by electroencephalography [EEG])

SECONDARY OUTCOMES:
Proportion of patients achieving electroclinical cessation of seizures | 12 hours
  Proportions of patients who achieve cessation of BOTH clinical seizures (as observed clinically) AND electrical seizures (evaluated by electroencephalography [EEG])
Time to electroclinical cessation of seizures | 24 hours
  Time to cessation of BOTH clinical seizures (as observed clinically) AND electrical seizures (evaluated by electroencephalography [EEG])
Proportion of patients achieving electroclinical seizure freedom | 24 hours
  Proportion of patients achieving freedom from BOTH clinical seizures (as observed clinically) AND electrical seizures (evaluated by electroencephalography [EEG])
Proportion of patients with super-refractory status epilepticus | 24 hours
  Proportion of patients with persistent seizures for 24 hours or more after initiation of 3rd line medications (anesthetics) or recurrence of seizure during withdrawal of the anesthetics
Proportion of patients with adverse gastrointestinal effects | 24 hours
  Proportion of patients with adverse gastrointestinal effects (vomiting, diarrhea, abdominal pain) evaluated by direct observation and patient-reporting
Change in blood beta-hydroxybutyrate level | From baseline to 30 minutes, 1 hour, 2 hours, 5 hours, 9 hours, and 12 hours study timepoints
  Change in blood level of beta-hydroxybutyrate
Change in blood glucose level | From baseline to 30 minutes, 1 hour, 2 hours, 5 hours, 9 hours, and 12 hours study timepoints
  Change in blood level of glucose
Change in blood pH | From baseline to 30 minutes, 1 hour, 2 hours, 5 hours, 9 hours, and 12 hours study timepoints
  Change in blood pH

OTHER OUTCOMES:
Change in blood bicarbonates level | From baseline to 30 minutes, 1 hour, 2 hours, 5 hours, 9 hours, and 12 hours study timepoints
  Change in blood bicarbonates level
Change in blood lactate level | From baseline to 30 minutes, 1 hour, 2 hours, 5 hours, 9 hours, and 12 hours study timepoints
  Change in blood lactate level
Change in hemoglobin level | From baseline to 1 hour and 12 hours study timepoints
  Change in hemoglobin level
Change in leukocyte count | From baseline to 1 hour and 12 hours study timepoints
  Change in leukocyte count
Change in platelets count | From baseline to 1 hour and 12 hours study timepoints
  Change in platelets count
Change in serum sodium level | From baseline to 1 hour and 12 hours study timepoints
  Change in serum sodium level
Change in serum potassium level | From baseline to 1 hour and 12 hours study timepoints
  Change in serum potassium level
Change in CRP level | From baseline to 1 hour and 12 hours study timepoints
  Change in CRP level
Change in lipid profile | From baseline to 1 hour and 12 hours study timepoints
  Change in lipid profile
Change in blood alanine transaminase level | From baseline to 1 hour and 12 hours study timepoints
  Change in blood alanine transaminase (ALT) level
Change in serum creatinine level | From baseline to 1 hour and 12 hours study timepoints
  Change in serum creatinine level

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrahim A Sadek, MD, PhD, Study Chair — Sohag University
Locations (1):
- Department of Pediatrics at Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Unidentified individual participant data (IPD) underlying study results will be available upon reasonable request
Supporting Information: Study Protocol, SAP
Time Frame: Unidentified individual participant data (IPD) underlying study results will be available upon reasonable request 6-months after publication

REFERENCES:
- [Background] Arya R, Peariso K, Gainza-Lein M, Harvey J, Bergin A, Brenton JN, Burrows BT, Glauser T, Goodkin HP, Lai YC, Mikati MA, Fernandez IS, Tchapyjnikov D, Wilfong AA, Williams K, Loddenkemper T; pediatric Status Epilepticus Research Group (pSERG). Efficacy and safety of ketogenic diet for treatment of pediatric convulsive refractory status epilepticus. Epilepsy Res. 2018 Aug;144:1-6. doi: 10.1016/j.eplepsyres.2018.04.012. Epub 2018 Apr 27. PMID 29727818
- [Background] Chomtho S, Uaariyapanichkul J, Chomtho K. Outcomes of parenteral vs enteral ketogenic diet in pediatric super-refractory status epilepticus. Seizure. 2022 Mar;96:79-85. doi: 10.1016/j.seizure.2022.01.019. Epub 2022 Feb 5. PMID 35158320
- [Background] Clarke K, Tchabanenko K, Pawlosky R, Carter E, Todd King M, Musa-Veloso K, Ho M, Roberts A, Robertson J, Vanitallie TB, Veech RL. Kinetics, safety and tolerability of (R)-3-hydroxybutyl (R)-3-hydroxybutyrate in healthy adult subjects. Regul Toxicol Pharmacol. 2012 Aug;63(3):401-8. doi: 10.1016/j.yrtph.2012.04.008. Epub 2012 May 3. PMID 22561291
- [Background] Gilbert DL, Pyzik PL, Freeman JM. The ketogenic diet: seizure control correlates better with serum beta-hydroxybutyrate than with urine ketones. J Child Neurol. 2000 Dec;15(12):787-90. doi: 10.1177/088307380001501203. PMID 11198492
- [Background] Schoeler NE, Simpson Z, Zhou R, Pujar S, Eltze C, Cross JH. Dietary Management of Children With Super-Refractory Status Epilepticus: A Systematic Review and Experience in a Single UK Tertiary Centre. Front Neurol. 2021 Mar 12;12:643105. doi: 10.3389/fneur.2021.643105. eCollection 2021. PMID 33776895
- [Background] Si J, Wang Y, Xu J, Wang J. Antiepileptic effects of exogenous beta-hydroxybutyrate on kainic acid-induced epilepsy. Exp Ther Med. 2020 Dec;20(6):177. doi: 10.3892/etm.2020.9307. Epub 2020 Oct 9. PMID 33101467
- [Background] Stubbs BJ, Cox PJ, Evans RD, Santer P, Miller JJ, Faull OK, Magor-Elliott S, Hiyama S, Stirling M, Clarke K. On the Metabolism of Exogenous Ketones in Humans. Front Physiol. 2017 Oct 30;8:848. doi: 10.3389/fphys.2017.00848. eCollection 2017. PMID 29163194
- [Background] Carson RP, Herber DL, Pan Z, Phibbs F, Key AP, Gouelle A, Ergish P, Armour EA, Patel S, Duis J. Nutritional Formulation for Patients with Angelman Syndrome: A Randomized, Double-Blind, Placebo-Controlled Study of Exogenous Ketones. J Nutr. 2021 Dec 3;151(12):3628-3636. doi: 10.1093/jn/nxab284. PMID 34510212
- [Background] Cox PJ, Kirk T, Ashmore T, Willerton K, Evans R, Smith A, Murray AJ, Stubbs B, West J, McLure SW, King MT, Dodd MS, Holloway C, Neubauer S, Drawer S, Veech RL, Griffin JL, Clarke K. Nutritional Ketosis Alters Fuel Preference and Thereby Endurance Performance in Athletes. Cell Metab. 2016 Aug 9;24(2):256-68. doi: 10.1016/j.cmet.2016.07.010. Epub 2016 Jul 27. PMID 27475046
- [Background] Trinka E, Cock H, Hesdorffer D, Rossetti AO, Scheffer IE, Shinnar S, Shorvon S, Lowenstein DH. A definition and classification of status epilepticus--Report of the ILAE Task Force on Classification of Status Epilepticus. Epilepsia. 2015 Oct;56(10):1515-23. doi: 10.1111/epi.13121. Epub 2015 Sep 4. PMID 26336950